CLINICAL TRIAL: NCT04825470
Title: Liver Transplantation in Patients With Unresectable GastroIntestinal Stromal Tumors (GIST) Liver Metastases
Brief Title: Liver Transplantation for Unresectable GIST Liver Metastases
Acronym: TRANSGIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Felipe Alconchel, MD, PhD, Principal Investigator, Hospital Universitario Virgen de la Arrixaca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRANSGIST
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Liver Diseases; Liver Cancer; Liver Metastases; Liver Neoplasms; Liver Mass; Liver Carcinoma; Liver Transplant; Complications; Liver Transplant Disorder; GIST; GIST, Malignant; Gastrointestinal Stromal Tumors; Gastrointestinal Stromal Tumor of Duodenum; Gastrointestinal Stromal Tumor of Rectum; Gastrointestinal Stromal Tumor of Other Sites; Gastrointestinal Stromal Tumor, Unspecified Site; Gastrointestinal Stromal Tumor of Stomach; Gastrointestinal Stromal Tumor of Esophagus (Disorder); Gastrointestinal Stromal Tumor by AJCC V8 Stage; Gastrointestinal Stromal Tumor, Malignant; Gastrointestinal Stromal Tumor (GIST) of the Gastrointestinal Tract; Gastrointestinal Stromal Tumor of Small Intestine (Disorder); Gastrointestinal Stromal Tumor of Large Intestine (Disorder); Metastases to Liver; Metastatic Liver Cancer; Metastasis; Metastases; Liver Transplantation; Transplant Oncology
Keywords: liver transplantation; gastrointestinal stromal tumor (GIST); Transplant Oncology; liver neoplasms; liver metastases
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms; Carcinoma, Hepatocellular; Gastrointestinal Stromal Tumors; Neoplasm Metastasis | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver Transplantation (Experimental)
  Interventions: Procedure: Liver Transplantation

INTERVENTIONS:
Procedure: Liver Transplantation — Liver Transplantation

SUMMARY:
Liver Transplantation for Unresectable GIST Liver Metastases

ELIGIBILITY:
Inclusion Criteria:

* GIST diagnosis (c-Kit, CD34, DOG-1)
* Imatinib-sensitive mutation
* Non-resectable liver metastases
* Abscence of extrahepatic disease
* Period greater than two years between primary tumor and metastases diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Through study completion, an average of 2 years
  Survival
Graft Survival | Through study completion, an average of 2 years
  Liver graft Survival

SECONDARY OUTCOMES:
Relapse free survival | Through study completion, an average of 2 years
Disease free survival | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Felipe Alconchel, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fernandez JA, Alconchel F, Gomez B, Martinez J, Ramirez P. Unresectable GIST liver metastases and liver transplantation: A review and theoretical basis for a new indication. Int J Surg. 2021 Oct;94:106126. doi: 10.1016/j.ijsu.2021.106126. Epub 2021 Sep 27. PMID 34592432
- See also: Research Registry — https://www.researchregistry.com/browse-the-registry#registryofsystematicreviewsmeta-analyses/registryofsystematicreviewsmeta-analysesdetails/606798f8d9bb31001bb1dab8/